CLINICAL TRIAL: NCT04976530
Title: Safe, Timely Antithrombotic Removal-Ticagrelor (STAR-T): Double-blind Randomized Study of Reduction in Bleeding by Ticagrelor Removal Via Intraop Use of DrugSorb-Antithrombotic Removal (ATR) in Cardiac Surgery Patients <2 Days of Drug Stop
Brief Title: Safe and Timely Antithrombotic Removal - Ticagrelor (STAR-T)
Acronym: STAR-T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CytoSorbents, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-01
Record Dates: First submitted 2021-07-06; First posted 2021-07-26 (Actual); Results first posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Hemorrhage, Surgical; Blood Loss, Surgical; Blood Loss, Postoperative; Hemorrhage Postoperative
MeSH Terms: conditions — Blood Loss, Surgical; Postoperative Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Control (Sham Comparator): Standard of care with Sham set-up
  Interventions: Device: Sham comparator
- DrugSorb-ATR Intervention (Experimental): Standard of care + DrugSorb-ATR system
  Interventions: Device: DrugSorb-ATR system

INTERVENTIONS:
Device: DrugSorb-ATR system — Sorbent hemoperfusion system integrated into the cardiopulmonary bypass (CPB) circuit
  Other Names: Sorbent hemoperfusion system
  Arms: DrugSorb-ATR Intervention
Device: Sham comparator — Sham comparator in similar position to the investigative device, but NOT integrated into the cardiopulmonary (CPB) circuit
  Arms: Control

SUMMARY:
Prospective, multi-center, double-blind, randomized pivotal trial to evaluate the safety and effectiveness of the DrugSorb-Antithrombotic Removal (ATR) system for intraoperative removal of ticagrelor in patients undergoing urgent cardiothoracic (CT) surgery with cardiopulmonary bypass (CPB).

DETAILED DESCRIPTION:
Antithrombotic agents such as ticagrelor can increase the risk of surgical bleeding in patients undergoing CT surgery if there is not adequate washout time of the drug. Patients who require urgent surgery may not be able to wait for the recommended washout time (up to 7 days). The intraoperative use of the DrugSorb-ATR device to remove active ticagrelor may help reduce the risk of postoperative surgical bleeding in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 years of age or older, with documented full, written informed consent
2. Requiring cardiothoracic (CT) surgery with cardiopulmonary bypass (CPB) within two days of ticagrelor discontinuation (day of last dose = day 0)

Exclusion Criteria:

1. CT surgery occurring 3 days or greater following ticagrelor discontinuation
2. Heart-lung transplant procedures
3. Procedures for implant or revision of left ventricular assist device (LVAD) or right ventricular assist device (RVAD)
4. Pre-existing conditions that pose a known risk for bleeding (i.e., heparin induced thrombocytopenia /thrombosis [HITT], perioperative platelet count < 50,000u/L, hemophilia, and international normalized ratio [INR] >1.5)
5. Prohibited concomitant antithrombotic medications as defined in the study protocol
6. Acute sickle cell crisis
7. Known allergy to device components
8. Active (untreated) systemic infection
9. History of major organ transplantation and those currently receiving immunosuppressive medication or who are profoundly immune suppressed
10. Women with positive pregnancy test during current admission or who are breast-feeding
11. Life expectancy <30 days
12. Inability to comply with requirements of the study protocol
13. Treatment with investigational drug or device within 30 days of current surgery
14. Previous enrollment in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Mack, MD, Principal Investigator — Baylor Scott & White The Heart Hospital; C. M Gibson, MD, Principal Investigator — Beth Israel Deaconess Medical Center, The Baim Institute, and Harvard Medical School; Richard Whitlock, MD, Principal Investigator — Hamilton General Hospital
Locations (29):
- United States (22):
  - University of California, Davis Medical Center, Sacramento, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - MedStar Health Research Institute, Washington D.C., District of Columbia
  - Emory University Hospital Midtown/Emory School of Medicine, Atlanta, Georgia
  - Lutheran Medical Group, Fort Wayne, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Mississippi, Jackson, Mississippi
  - Virtua Health, Marlton, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - New York University Langone Health, New York, New York
  - University Hospitals, Cleveland Medical Center, Cleveland, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor Scott & White The Heart Hospital Plano, Plano, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - VCU Medical Center, Richmond, Virginia
  - Carilion Clinic, Roanoke, Virginia
  - University of Wisconsin-Madison, Madison, Wisconsin
  - The Medical College of Wisconsin, Inc., Milwaukee, Wisconsin
- Canada (7):
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Hamilton General Hospital, Hamilton Health Sciences Corporation, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Health Sciences Centre, University Hospital, London, Ontario
  - St. Michael's Hospital, Unity Health Toronto, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec - Université Laval, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mould DR, Sweeney KR, Prats J, Fan W, Schneider DJ, Storey RF, Deliargyris EN. Pharmacokinetic Modeling of Ticagrelor and Ticagrelor Active Metabolite Removal by the DrugSorb-ATR Device in a Randomized Controlled Study of Patients Undergoing Cardiac Surgery. J Cardiovasc Pharmacol. 2026 Feb 1;87(2):105-113. doi: 10.1097/FJC.0000000000001779. PMID 41642317
- [Derived] Tripathi R, Morales J, Lee V, Gibson CM, Mack MJ, Schneider DJ, Douketis J, Sellke FW, Ohman ME, Thourani VH, Storey RF, Deliargyris EN. Antithrombotic drug removal from whole blood using Haemoadsorption with a porous polymer bead sorbent. Eur Heart J Cardiovasc Pharmacother. 2022 Dec 2;8(8):847-856. doi: 10.1093/ehjcvp/pvac036. PMID 35657375

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | DrugSorb-ATR Intervention
Started | 70 | 70
Completed | 70 | 70
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population = modified intent to treat (mITT), ie, randomized subjects who had surgery and received a study device (control or intervention).
Groups:
- DrugSorb-ATR Intervention: Standard of care + DrugSorb-ATR system
  DrugSorb-Antithrombotic Removal (ATR) system: Sorbent hemoperfusion system integrated into the cardiopulmonary bypass (CPB) circuit
- Total: Total of all reporting groups
Arm/Group | Control | DrugSorb-ATR Intervention | Total
Number analyzed (Participants) | 66 | 66 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (8.54) | 64.4 (10.63) | 64.5 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 56 | 56 | 112
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 50 | 53 | 103
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 6 | 11
Region of Enrollment [Number; unit: participants]
  Canada | 22 | 23 | 45
  United States | 44 | 43 | 87
Hypertension [Count of Participants; unit: Participants] | 58 | 54 | 112
Heart failure [Count of Participants; unit: Participants] | 23 | 18 | 41
Coronary artery disease [Count of Participants; unit: Participants] | 62 | 61 | 123
Thrombocytopenia [Count of Participants; unit: Participants] | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Perioperative (Periop) Bleeding, Primary Effectiveness Composite Endpoint, Modified Intent to Treat (mITT) Population
Description: Incidence of periop bleeding, primary effectiveness composite endpoint, mITT population. Primary effectiveness endpoint was a composite of (ranked) 1) fatal periop bleeding; 2) moderate, severe, or massive bleeding events based on the universal definition for periop bleeding (UDPB) >2 classification; and 3) 24 hour chest tube drainage (CTD) volume; evaluated by an unmatched win ratio method. Using the hierarchical order of the components of each composite endpoint every patient in the Sham arm is compared with every patient in the DrugSorb-ATR arm to make Ns x Nd pairs. The numbers below are the number of 'winners' for two treatments; 'win' is given for the better outcome in the pair, eg, less bleeding. The win ratio is the total number of winners in DrugSorb-ATR arm divided by the total number of winners in Sham arm. A ratio of wins > 1.0 favors the treatment arm. 95% confidence interval (CI) and p-value are calculated accordingly. The win ratio is 1.07 (95% CI 0.72, 1.58), p=0.748.
Time Frame: Through the first 48hrs post-operation
Population: mITT, modified intent-to-treat
Measure: Number; unit: number of wins
Arm/Group | Control | DrugSorb-ATR Intervention
Number analyzed (Participants) | 66 | 66
number of wins | 2103 | 2244
Statistical Analysis 1: Comparison: Control vs DrugSorb-ATR Intervention; Test type: Superiority; p = 0.748, Finkelstein Schoenfeld test; win ratio = 1.07, 95% CI 2-sided [0.72 to 1.58]

2. Primary Outcome: Incidence of Perioperative (Periop) Bleeding, Primary Effectiveness Composite Endpoint, Isolated Coronary Artery Bypass Grafting (I-CABG) Per Protocol (PP) Population
Description: Incidence of periop bleeding, primary effectiveness composite endpoint, i--CABG population. The primary effectiveness endpoint was a composite of (ranked) 1) fatal periop bleeding; 2) moderate, severe, or massive bleeding events based on the universal definition for periop bleeding (UDPB) >2 classification; and 3) 24 hour chest tube drainage (CTD) volume; evaluated by an unmatched win ratio method. Using the hierarchical order of the components of each composite endpoint every patient in the Sham arm is compared with every patient in the DrugSorb-ATR arm to make Ns x Nd pairs. The numbers below are the number of 'winners' for two treatments; 'win' is given for the better outcome in the pair, eg, less bleeding. The win ratio is the total number of winners in DrugSorb-ATR arm divided by the total number of winners in the Sham arm. A ratio of wins >1.0 favors the treatment arm. The win ratio was 1.33 (95% confidence interval 0.86, 2.04) p-value 0.202.
Time Frame: Through the first 48hrs post operation
Population: i-CABG, isolated CABG, per protocol population
Measure: Number; unit: number of wins
Arm/Group | Control | DrugSorb-ATR Intervention
Number analyzed (Participants) | 60 | 51
number of wins | 1310 | 1741
Statistical Analysis 1: Comparison: Control vs DrugSorb-ATR Intervention; Test type: Superiority; p = 0.202, Finkelstein Schoenfeld test; win ratio = 1.33, 95% CI 2-sided [0.86 to 2.04]

3. Primary Outcome: Incidence of Perioperative (Periop) Bleeding, Supplemental Primary Effectiveness Composite Endpoint, mITT Population
Description: Incidence of Periop Bleeding, Supplemental Primary Effectiveness Composite Endpoint, mITT population. The supplementary primary effectiveness endpoint was a composite of (ranked) 1) fatal periop bleeding; 2) severe, or massive bleeding events based on the universal definition for periop bleeding (UDPB) >3 classification; and 3) 24 hour chest tube drainage (CTD) volume; evaluated by an unmatched win ratio method. Using the hierarchical order of the components of each composite endpoint every patient in the Sham arm is compared with every patient in the DrugSorb-ATR arm to make Ns x Nd pairs. The numbers given below are the number of 'winners' for two treatments; a 'win' is given for the better outcome in the pair, eg, less bleeding. The win ratio is the total number of winners in DrugSorb-ATR arm divided by the total number of winners in Sham arm. A ratio of wins >1.0 favors the treatment arm. The win ratio was 1.17 (95% confidence interval 0.79, 1.73) p value 0.451.
Time Frame: Through the first 48 hours post-operation
Population: mITT, modified intent-to-treat
Measure: Number; unit: number of wins
Arm/Group | Control | DrugSorb-ATR Intervention
Number analyzed (Participants) | 66 | 66
number of wins | 2005 | 2336
Statistical Analysis 1: Comparison: Control vs DrugSorb-ATR Intervention; Test type: Superiority; p = 0.451, Finkelstein Schoenfeld test; win ratio = 1.17, 95% CI 2-sided [0.79 to 1.73]

4. Primary Outcome: Incidence of Perioperative (Periop) Bleeding, Supplemental Primary Effectiveness Composite Endpoint, I-CABG Per Protocol (PP) Population
Description: Incidence of Periop Bleeding, Supplemental Primary Effectiveness Composite Endpoint, I-CABG population. The supplementary primary effectiveness endpoint was a composite of (ranked) 1) fatal periop bleeding; 2) severe, or massive bleeding events based on the universal definition for periop bleeding (UDPB) >3 classification; and 3) 24 hour chest tube drainage (CTD) volume; evaluated by an unmatched win ratio method. Using the hierarchical order of the components of each composite endpoint every patient in the Sham arm is compared with every patient in the DrugSorb-ATR arm to make Ns x Nd pairs. The numbers below are the number of 'winners' for two treatments; a 'win' is given for the better outcome in the pair, eg, less bleeding. The win ratio is the total number of winners in DrugSorb-ATR arm divided by the total number of winners in Sham arm. A ratio of wins >1.0 favors the treatment arm. The win ratio was 1.59 (95% confidence interval 1.02, 2.46) p-value 0.041.
Time Frame: Through the first 48hrs post-operation
Population: i-CABG PP: subjects undergoing isolated CABG procedures, per protocol (those without major protocol deviations that would affect determination of device effectiveness.
Measure: Number; unit: number of wins
Arm/Group | Control | DrugSorb-ATR Intervention
Number analyzed (Participants) | 60 | 51
number of wins | 1178 | 1868
Statistical Analysis 1: Comparison: Control vs DrugSorb-ATR Intervention; Test type: Superiority; p = 0.041, Finkelstein Schoenfeld test; win ratio = 1.59, 95% CI 2-sided [1.02 to 2.46]

5. Secondary Outcome: Chest Tube Drainage, mITT Population
Description: Drainage volume from all chest and mediastinal tubes
Time Frame: Through 24hrs post-operation
Population: mITT (all enrolled subjects who received a study device)
Measure: Median (Full Range); unit: mL
Arm/Group | Control | DrugSorb-ATR Intervention
Number analyzed (Participants) | 66 | 66
mL | 746 [200 to 2670] | 715 [205 to 8956]
Statistical Analysis 1: Comparison: Control vs DrugSorb-ATR Intervention; Test type: Superiority; p = 0.6, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Chest Tube Drainage, i-CABG PP Population
Description: Drainage volume from all chest and mediastinal tubes
Time Frame: Through 24hrs post-operation
Population: isolated CABG per protocol population
Measure: Median (Full Range); unit: mL
Arm/Group | Control | DrugSorb-ATR Intervention
Number analyzed (Participants) | 60 | 51
mL | 765 [200 to 2670] | 645 [205 to 3425]
Statistical Analysis 1: Comparison: Control vs DrugSorb-ATR Intervention; Test type: Superiority; p = 0.079, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Chest Tube Drainage, mITT Population
Description: Drainage volume from all chest and mediastinal tubes
Time Frame: Through 12hrs post-operation
Population: mITT (all enrolled subjects who received a study device)
Measure: Median (Full Range); unit: mL
Arm/Group | Control | DrugSorb-ATR Intervention
Number analyzed (Participants) | 66 | 66
mL | 487 [140 to 1690] | 430 [35 to 8050]
Statistical Analysis 1: Comparison: Control vs DrugSorb-ATR Intervention; Test type: Superiority; p = 0.427, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Chest Tube Drainage, i-CABG PP Population
Description: Drainage volume from all chest and mediastinal tubes
Time Frame: Through 12hrs post-operation
Population: isolated CABG per protocol population
Measure: Median (Full Range); unit: mL
Arm/Group | Control | DrugSorb-ATR Intervention
Number analyzed (Participants) | 60 | 51
mL | 487 [165 to 1690] | 410 [35 to 1480]
Statistical Analysis 1: Comparison: Control vs DrugSorb-ATR Intervention; Test type: Superiority; p = 0.042, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Packed Red Blood Cell (PRBC) Transfusions (Units), mITT Population
Description: Total PRBC transfusions (units) during hospitalization in the mITT population
Time Frame: From procedure start through to discharge from index hospitalization, on average 1-2 weeks
Population: mITT
Measure: Median (Full Range); unit: PBRC Units
Arm/Group | Control | DrugSorb-ATR Intervention
Number analyzed (Participants) | 35 | 40
PBRC Units | 3 [1 to 10] | 2.5 [1 to 25]

10. Secondary Outcome: PRBC Transfusions, (Units) I-CABG PP Population
Description: Total PRBC transfusions (units) during hospitalization
Time Frame: From procedure start through to discharge from index hospitalization, on average 1-2 weeks
Population: I-CABG PP, isolated CABG per protocol population
Measure: Median (Full Range); unit: PRBC units
Arm/Group | Control | DrugSorb-ATR Intervention
Number analyzed (Participants) | 30 | 27
PRBC units | 3 [1 to 10] | 2 [1 to 20]

11. Secondary Outcome: Platelet Transfusions (Units), mITT Population
Description: Total Platelet transfusions (units) during hospitalization
Time Frame: From procedure start through to discharge from index hospitalization, on average 1-2 weeks
Population: mITT
Measure: Median (Full Range); unit: PBRC units
Arm/Group | Control | DrugSorb-ATR Intervention
Number analyzed (Participants) | 27 | 31
PBRC units | 2 [1 to 5] | 2 [1 to 10]

12. Secondary Outcome: Platelet Transfusions, (Units), I-CABG PP Population
Description: Total Platelet transfusions (units) during hospitalization
Time Frame: From procedure start through to discharge from index hospitalization, on average 1-2 weeks
Population: I-CABG PP, isolated CABG per protocol population
Measure: Median (Full Range); unit: Platelet units
Arm/Group | Control | DrugSorb-ATR Intervention
Number analyzed (Participants) | 24 | 21
Platelet units | 2 [1 to 5] | 2 [1 to 8]

ADVERSE EVENTS:
Time Frame: 30 days
Description: The primary safety endpoint of this study was to evaluate the product safety profile through the Good Clinical Practice level assessment of adverse events (AEs) during the study period. This study evaluated a device, therefore, in this section we report all Device-related serious adverse events (SAEs).
Arm/Group | Control | DrugSorb-ATR Intervention
All-Cause Mortality (participants affected / at risk) | 1/66 | 1/66
Serious Adverse Events (participants affected / at risk) | 19/66 | 25/66
Other Adverse Events (participants affected / at risk) | 57/66 | 58/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=66) | DrugSorb-ATR Intervention (N=66)
Atrial fibrillation (Cardiac disorders) | 4 | 0
Cardiac tamponade (Cardiac disorders) | 3 | 0
Cardiogenic shock (Cardiac disorders) | 2 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Right ventricular failure (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Ventricular dysfunction (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 3
Coagulopathy (Blood and lymphatic system disorders) | 0 | 2
Blood loss anaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 3
Haemorrhage (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Shock haemorrhage (Vascular disorders) | 0 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 2 | 0
Vasoplegia syndrome (Injury, poisoning and procedural complications) | 2 | 0
Post-procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Cerebral vascular event (Nervous system disorders) | 0 | 3
Lacunar infarction (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Medical device site haemorrhage (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Paravalvular regurgitation (General disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 3
Gout (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic alkalosis (Metabolism and nutrition disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
International normalized ratio increased (Investigations) | 1 | 0
Device breakage (Product Issues) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=66) | DrugSorb-ATR Intervention (N=66)
Atrial fibrillation (Cardiac disorders) | 22 | 28
Pericarditis (Cardiac disorders) | 4 | 2
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 13 | 16
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Anaemia (Blood and lymphatic system disorders) | 11 | 11
Leukocytosis (Blood and lymphatic system disorders) | 5 | 7
Blood loss anaemia (Blood and lymphatic system disorders) | 8 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 8
Hypotension (Vascular disorders) | 6 | 9
Investigations (Vascular disorders) | 10 | 12
Blood albumin decreased (Vascular disorders) | 2 | 5
Protein total decreased (Vascular disorders) | 2 | 4
Procedural pain (Injury, poisoning and procedural complications) | 4 | 3
Vasoplegia syndrome (Injury, poisoning and procedural complications) | 5 | 2
Anemia postoperative (Injury, poisoning and procedural complications) | 1 | 4
Acute kidney injury (Renal and urinary disorders) | 3 | 12
General disorders and administration site conditions (Renal and urinary disorders) | 8 | 10
Oedema peripheral (Renal and urinary disorders) | 2 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 4
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 5
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 1
Gastrointestinal disorders (Gastrointestinal disorders) | 7 | 9
Constipation (Gastrointestinal disorders) | 4 | 5
Psychiatric disorders (Psychiatric disorders) | 2 | 7
Delirium (Psychiatric disorders) | 0 | 5

LIMITATIONS AND CAVEATS:
Ticagrelor blood levels comprise 99.8% protein-bound drug and 0.2% free, pharmacologically active drug. The device removes free ticagrelor and blood samples were collected during the study to assess reduction in free ticagrelor levels as a secondary endpoint. However, an assay that measures free ticagrelor is not commercially available and therefore data for free drug removal was not collected in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-05-26): https://cdn.clinicaltrials.gov/large-docs/30/NCT04976530/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-24): https://cdn.clinicaltrials.gov/large-docs/30/NCT04976530/SAP_001.pdf